CLINICAL TRIAL: NCT04059367
Title: An Open-label, Single-sequence, Crossover Trial Investigating the Influence of NNC9204-1177 on Pharmacokinetics of Index Substrates for Cytochrome P450 Enzymes
Brief Title: Research Study to Investigate How a Study Medicine (NNC9204- 1177) Affects Blood Levels of Other Medicines in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9277-4555; U1111-1232-7100 Trial (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Single-sequence, cross-over drug interaction trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNC9204-1177 and cocktail of approved drugs (Experimental)
  Interventions: Drug: NNC9204-1177; Drug: Cocktail of 5 already approved drugs

INTERVENTIONS:
Drug: NNC9204-1177 — Increasing doses of NNC9204-1177 administered s.c. (subcutaneously, under the skin) in the stomach area once-weekly for 11 weeks
Drug: Cocktail of 5 already approved drugs — 5 medicines as tablets, capsules or syrup to be taken with water on Day 1 and Day 78 of the study

SUMMARY:
The study looks at how the study medicine (NNC9204-1177) affects other medicines in the body. Participants will get the study medicine and 5 other medicines which have all been approved by the authorities. Participants will get 1 injection of the study medicine each week for 11 weeks. The study medicine is injected under the skin in the stomach area. All injections will be given by study staff. Participants will get 5 medicines as tablets, capsules or syrup to be taken with water at the beginning of the study and after 10 weeks of treatment with the study medicine. The study will last for about 4 months. Participants will have 14 visits to the clinic with the study staff and study doctor. Participants will have blood draws and 2 different kinds of electrocardiograms taken during the study. They will be asked about your mental health. People who use any medication, including herbal products, cannot take part in the study. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period or if they use birth control pills or other hormonal birth control products.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-60 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 23.0 and 29.9 kg/m^2 (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method (intra-uterine device (IUD), vasectomised partner or sexual abstinence)
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs, except for IUDs, within 14 days prior to the day of screening.
* Use of any herbal medicine known to interfere with the metabolic CYP pathways, such as Hypericum (St. John's Wort), ginseng, garlic, milk thistle, and echinaceae, within 14 days prior to the day of screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve extrapolated to infinity of the caffeine | From 0 to 24 hours after a single dose of caffeine without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng*h/mL
Area under the plasma concentration-time curve extrapolated to infinity of the omeprazole | From 0 to 8 hours after a single dose of omeprazole without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng*h/mL
Area under the plasma concentration-time curve extrapolated to infinity of the midazolam | From 0 to 12 hours after a single dose of midazolam without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng*h/mL
Area under the plasma concentration-time curve extrapolated to infinity of the s-warfarin | From 0 to 168 hours after a single dose of warfarin without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng*h/mL
Area under the plasma concentration-time curve extrapolated to infinity of the dextromethorphan | From 0 to 72 hours after a single dose of dextromethorphan without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng*h/mL

SECONDARY OUTCOMES:
Maximum observed plasma caffeine concentration after a single dose | From 0 to 24 hours after a single dose of caffeine without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng/mL
Maximum observed plasma omeprazole concentration after a single dose | From 0 to 8 hours after a single dose of omeprazole without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng/mL
Maximum observed plasma s-warfarin concentration after a single dose | From 0 to 168 hours after a single dose of warfarin without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng/mL
Maximum observed plasma midazolam concentration after a single dose | From 0 to 12 hours after a single dose of midazolam without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng/mL
Maximum observed plasma dextromethorphan concentration after a single dose | From 0 to 72 hours after a single dose of dextromethorphan without NNC9204-1177 exposure (administered on Visit 2, Day 1) and at NNC9204-1177 steady state (administered on Visit 12, Day 78)
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com